CLINICAL TRIAL: NCT06684899
Title: An In-depth Appraisal of Cytokine-induced Killer Cells in Glioblastomas Patients
Brief Title: Optimizing Cytokine-Induced Killer Cells in Glioblastoma Patients
Acronym: KillGlio
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Giacomo Sferruzza, Principal Investigator, IRCCS San Raffaele
Other Study IDs: KillGlio
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Glioblastoma; Cytokine-Induced Killer Cells
Keywords: Glioblastoma; Cytokine-Induced Killer Cells
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients affected by glioblastoma: Subject with a documented diagnosis of glioblastoma (WHO criteria 2021), as confirmed by reference histopathology at San Raffaele Hospital.
- Healthy controls: Healthy donors will also be enrolled in the study to serve as controls in the manufacturing process and exploratory analysis. They will be recruited among healthy individuals attending our Unit

SUMMARY:
The goal of this prospective observational cohort study is to assess the optimal in vitro production protocol for generating Cytokine-Induced Killer (CIK) cells, a type of T lymphocyte, and to evaluate the potential adverse effects of concurrent neuro-oncology therapies on these cells in glioblastoma (GBM) patients. Additionally, the study aims to explore mechanisms to enhance the antitumor activity of CIK cells against GBM by investigating GBM's immune escape mechanisms that may counteract the Human Leukocyte Antigen (HLA)-independent activity of CIK cells.

The main questions it aims to answer are:

What is the most effective in vitro production protocol for generating highly active CIK cells from GBM patients? Do concurrent chemoradiotherapy or steroid treatments interfere with the activation or efficacy of CIK cells? What are potential strategies to counteract GBM immune escape mechanisms against CIK cells? Researchers will compare CIK cells produced under different protocols, including the use of media supplemented with commercial blood derivatives, to identify the most effective protocol and evaluate the impact of concomitant therapies on CIK cell functionality.

Participants will:

Undergo a single peripheral blood collection (GBM patients and healthy controls).

Have mononuclear cells isolated from their blood samples and expanded in vitro as CIK cells using various production protocols.

Have their CIK cells tested in vitro to assess activation status and antitumor activity, identifying optimal production methods and potential strategies to overcome GBM immune escape.

DETAILED DESCRIPTION:
The aim of this study is to optimize the expansion and manufacturing protocol of CIK cells obtained from patients with glioblastoma (GBM) and to assess their interaction with clinical variables, including the use of concomitant steroid therapy and alkylating chemotherapy. The study addresses multiple hypotheses, each corresponding to a specific aim of the project.

For the manufacturing process optimization, the primary hypothesis is that adding hemoderivatives (such as commercial human serum or platelet-derived lysate) can enhance the efficiency of Cytokine-Induced Killer (CIK) cell production (primary endpoint: higher fold expansion) and improve the quality of the final cell product (secondary endpoint: higher CIK viability and anticancer activity). This hypothesis is supported by published data but has not been tested on CIK cells expanded from GBM patients.

The second aim of the study is to evaluate the potential adverse effects of commonly used neuro-oncology therapies on CIK cells. Specifically, the investigators hypothesize that steroids, like dexamethasone, may have a detrimental effect by exerting cytotoxicity and reducing the anticancer activity of CIK cells. Although this hypothesis has been demonstrated for other lymphocyte types, it has not been explored for CIK cells. Establishing potential thresholds for toxicity (median toxic dose) could provide valuable information beyond neuro-oncology applications, considering the broad use of CIK cells in treating hematologic and solid tumors.

Additionally, the study will examine the potential negative impact of temozolomide on CIK therapy. Temozolomide, an alkylating agent, has shown differential cytotoxicity for lymphocytes, with T cells being more sensitive than Natural Killer (NK) cells. The hypothesis here is that CIK cells may inherit the sensitivity to temozolomide from their CD3+ T cell origins. This is particularly relevant, as a recent multicenter Phase III clinical trial evaluating CIK therapy in GBM scheduled CIK cell infusions to coincide with the adjuvant phase of the standard regimen, which involves a higher dosage of temozolomide.

The second part of the study will focus on exploring the immune escape mechanisms employed by GBM to evade Human Leukocyte Antigen (HLA)-independent immunosurveillance, like that mediated by CIK cells.

To achieve these aims, GBM patients will be enrolled at San Raffaele Hospital prior to the start of radiochemotherapy, along with healthy donors (HDs) as controls. Each participant will provide a single peripheral blood sample (approximately 10 ml) in an ethylenediaminetetraacetic acid (EDTA) tube. The study is designed as a cross-sectional study with a single time point for biological sample collection. Approximately 40 participants (20 patients and 20 healthy volunteers) will be enrolled over a 24-month period, allowing us to target Aim 1 (5 patients and 5 HDs), Aim 2 (5 patients and 5 HDs), and the exploratory analysis (10 patients and 10 HDs). An additional non-recruitment period of 12 months is planned for data analysis and manuscript preparation.

Epidemiological data will be collected for all subjects, including age, sex, relevant comorbidities, and medication usage. For GBM patients, additional oncological history details will be recorded, including steroid use (yes/no, dosage, and timing) and surgical treatment timing.

Following blood collection, Peripheral Blood Mononuclear Cells (PBMCs) will be isolated by Ficoll gradient centrifugation and expanded in vitro for 21 days, with sequential treatments of IFN-γ, OKT3, and Interleukin-2 (IL-2). Cells will be manually counted using trypan blue dye, and their phenotype will be characterized by flow cytometry. The anticancer activity of CIK cells will be assessed by co-culturing them with glioma cells and evaluating their degranulation ability (CD107a assay) and cytotoxic activity against target cells, as detected by flow cytometry.

ELIGIBILITY:
Inclusion Criteria for the glioblastoma (GBM) cohort:

* Age ≥18 years.
* Subject is willing and able to provide informed consent for participation in the study.
* Subject with a documented diagnosis of GBM (WHO criteria 2021), as confirmed by reference histopathology at San Raffaele Hospital.

Inclusion Criteria for the Healthy Volunteer Cohort:

* Age ≥18 years.
* Subject is willing and able to provide informed consent for participation in the study.
* Subjects In good general health as evidenced by medical history

Exclusion Criteria:

* Subject is not willing or able to provide informed consent for participation in the study. - Pregnancy
* Presence of an acute infection requiring active treatment.
* Documented ematological abnormalities: leukocytes < 3,000/μl or lymphocytes < 500/μl or neutrophils < 1,000/μl or hemoglobin < 9 g/100 ml or thrombocytes < 100,000/μl, based on the most recent laboratory tests performed for clinical practice.
* Documented immune deficiency
* Documented autoimmune disease.
* Documented positive serology for HIV or HBs antigen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will screen the patients affected by glioblastoma, diagnosed at the San Raffaele Hospital according to the World Health Organization criteria 2021. Patients fulfilling the inclusion and exclusion criteria will be enrolled and a blood sample will be obtained in the window period between the diagnosis (biopsy or tumor debulking) and the start of the standard radio-chemotherapy regimen. Both male and female patients will be enrolled to obtain, if possible, equal representation in the analysis.
  Healthy donors will also be enrolled in the study to serve as controls in the manufacturing process and exploratory analysis.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
To optimize the manufacturing process to obtain CIK from patients affected by GBM. | From 3 to 5 weeks after enrollment
  Cytokine-induced killer cells will be expanded from patients affected by glioblastoma according to different protocols. A statistically significant higher expansion fold compared to the standard (serum-free) protocol will be considered the primary endpoint of Aim 1
To establish the best applicability conditions of CIK in patients affected by GBM. | From 3 to 5 weeks after enrollment
  Cytokine-induced killer (CIK) cells will be treated with sequential doses of dexamethasone and temozolomide. The determination of the median toxic dose (TD50) will be considered as the endpoint to explore the concomitant use of these therapies.

IPD SHARING:
Plan to Share IPD: No